CLINICAL TRIAL: NCT01757236
Title: Prospective,Randomized,Open Label,European Multicenter Study of the Efficacy of the Linezolid-rifampin Combination Versus Standard of Care in the Treatment of Gram-positive.
Brief Title: Efficacy and Safety Study of Antibiotic Treatment to Treat Hip Prosthetic Joint Infection
Acronym: LIZ-BONE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: Pfizer (Industry); International Clinical Trials Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHAO2011/LB/LIZ-BONE; 2012-000781-38 (EudraCT Number)
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Hip Prosthetic Joint Infection
Keywords: Antibiotic; linezolid; linezolid/rifampin
MeSH Terms: interventions — Vancomycin; Ceftriaxone; Clindamycin; Sulfamethoxazole; Trimethoprim; Trimethoprim, Sulfamethoxazole Drug Combination; Fluoroquinolones; Linezolid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment A (Active Comparator): IV vancomycin (15mg/kg every 12 hours or in a continuous infusion) and IV ceftriaxone (2g daily) until Day 2 to 7 (until the susceptibility test results are obtained).
  Patients with only a confirmed Gram-positive infection will continue the study and will receive standard of care antibiotic therapy including oral rifampin (10-15mg/kg every 12 hours) combined with either oral clindamycin (600 mg every 8 hours) or oral sulfamethoxazole and trimethoprim (800/160 mg every 8 hours) or oral fluoroquinolone (Ofloxacin 200 mg every 12 hours). The total duration of antibiotic therapy from the day of the surgical procedure until the end of treatment (EOT) will be 6 weeks.
  Interventions: Drug: VANCOMYCIN; Drug: CEFTRIAXONE; Drug: CLINDAMYCIN; Drug: SULFAMETHOXAZOLE AND TRIMETHOPRIM (CO-TRIMOXAZOLE); Drug: FLUOROQUINOLONE; Drug: RIFAMPIN
- Treatment B (Experimental): IV vancomycin (15mg/kg every 12 hours or in a continuous infusion) and IV ceftriaxone (2g daily) until Day 2 to 7 (until the susceptibility test results are obtained).
  Patients with only a confirmed Gram-positive infection will continue the study and will receive oral linezolid (600mg every 12 hours) combined with oral rifampin (10-15mg/kg every 12 hours).
  The total duration of antibiotic therapy from the day of the surgical procedure until the end of treatment (EOT) will be 6 weeks.
  Interventions: Drug: VANCOMYCIN; Drug: CEFTRIAXONE; Drug: LINEZOLID; Drug: RIFAMPIN
- Treatment C (Experimental): IV linezolid (600 mg every 12 hours)and IV ceftriaxone (2g daily) until Day 2. Oral or IV rifampin (10-15 mg/kg every 12 hours) will be added 48 hours after initiating the study treatment. Treatment with the study drug will continue until Day 2 to 7 (until the susceptibility test results are obtained). Patients with only a confirmed Gram-positive infection will continue the study. Treatment with ceftriaxone will be discontinued and the patient will switch to oral linezolid and oral rifampin. The total duration of antibiotic therapy from the day of the surgical procedure until the end of treatment (EOT) will be 4 weeks.
  Interventions: Drug: VANCOMYCIN; Drug: CEFTRIAXONE; Drug: LINEZOLID; Drug: RIFAMPIN

INTERVENTIONS:
Drug: VANCOMYCIN
  Other Names: VANCOCIN
Drug: CEFTRIAXONE
  Other Names: ROCEPHIN
Drug: CLINDAMYCIN
  Other Names: DALACIN
  Arms: Treatment A
Drug: SULFAMETHOXAZOLE AND TRIMETHOPRIM (CO-TRIMOXAZOLE)
  Other Names: BACTRIM
  Arms: Treatment A
Drug: FLUOROQUINOLONE
  Other Names: OFLOCIN
  Arms: Treatment A
Drug: LINEZOLID
  Other Names: ZYVOXID
  Arms: Treatment B; Treatment C
Drug: RIFAMPIN
  Other Names: RIFADIN

SUMMARY:
The purpose of this study is to evaluate the efficacy of oral linezolid-rifampin combination therapy (over 4 or 6 weeks) versus the standard of care in the treatment of Gram-positive prosthetic hip joint infection with a one-stage surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 to ≤ 80 years of age, weight ≥ 40 kg, BMI < 35, who have received a diagnosis of chronic PJI (lasting more than 4 weeks but less than 24 months) requiring a one-stage surgical procedure and presenting at least ONE of the following clinical signs and symptoms:

   1. Joint pain
   2. Effusion
   3. Erythema and sensation of heat at the implant site
   4. Limited range of motion in the affected joint
2. Intraoperative microbiological specimens: during the surgical resection, 5 separate surgical specimens (at least 3) must be sent for culture and susceptibility testing. These specimens must be taken from different locations such as: Hip capsule, femoral membrane, acetabular membrane, synovium, and synovial fluid with separate instruments. A minimum of 2 surgical specimens must be positive. If a preoperative puncture revealed the presence of an acceptable (Gram+) pathogen, it is acceptable if only one pathogen similar to the previously revealed one is identified during the surgical procedure.
3. Documented presence of Gram-positive bacteria as sole pathogen responsible for the infection.

   Note: This criterion must be verified after obtaining the results of the susceptibility test performed on the specimens taken during the surgical procedure. The verification will occur between Day 2 and Day 7 of the study.
4. All patients must undergo 1-stage revision surgery.
5. IRB or IEC approved informed consent form signed and dated. Informed consent will be obtained from each patient before participation in this research study. If any patient is unable to give consent, it may be obtained from the patient's next of kin or legal representative in accordance with current laws and regulations.
6. Willing and able to comply with scheduled visits, up to 6 weeks of treatment with the study antibiotics, laboratory tests, and other study procedures.
7. Patient entitled to Health System benefits or other such benefits

Exclusion Criteria:

1. Concerning women of childbearing age:

   1. intake of oral contraceptives (estroprogestins and progestins)
   2. unability to use adequate mechanical contraceptive precautions
   3. a positive pregnancy test result within 72 hours prior to randomization
   4. pregnant, or are currently breastfeeding and unwilling to discontinue breastfeeding during therapy
2. Patients with a prosthetic joint infection caused by: Gram-negative, mixed Gram-negative and Gram-positive, fungal, or mycobacterial microorganisms. If a previous radiologically guided puncture has revealed the presence of a Gram-negative microorganism, the patient must not be enrolled in this study.
3. Platelet count less than 100 ×103/mm3 at the time of the examination performed during the screening period.
4. Hemoglobin < 9 g/dL at the time of the examination performed during the screening period.
5. Infection affecting several joints.
6. Rheumatological disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.)
7. Previously diagnosed immune function disease(s) (e.g., AIDS), neutropenia (neutrophils < 1000/mm3).
8. Alcoholism or substance abuse sufficient, in the investigator's judgment, to prevent treatment adherence to the study drug and/or follow-up.
9. Patients currently in peritoneal dialysis or receiving another treatment for renal failure (e.g., hemofiltration, CVVH).
10. Liver failure with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) and/or total bilirubin levels upper or egal to 5 times the upper limit of normal.
11. Patients with other concurrent serious infections such as: endocarditis, meningitis, or central nervous system (CNS) infections, decubitus and ischemic ulcers with underlying osteomyelitis, necrotizing fasciitis, gas gangrene. If suspected, these diagnoses must be ruled out prior to enrollment in the study.
12. Previous randomization in this protocol.
13. Not expected or not likely to survive for the entire duration of the treatment period and TOC (12 months after the end of treatment).
14. Hypersensitivity to the study drugs or their excipients.
15. Identification of a pathogen resistant to the investigational drugs.
16. Patients treated with a protease inhibitor(e.g. indinavir, ritonavir), or with delavirdine, or with nevirapine.
17. Patients treated or having been treated within two weeks prior surgery with an MAOI (A or B), an antiserotonergic drug, a tricyclic antidepressant, an agonist of 5HT1-receptor(triptan), a direct or indirect sympathomimetic drug (including adrenergic bronchodilator, pseudoephedrin, phenylpropanolamin), a vasopressor (adrenalin, noradrenalin), dopaminergic drug, pethidin or buspirone,
18. Patients with a degenerative neurological disease (Parkinson's disease, multiple sclerosis, Alzheimer's disease, etc.).
19. Patient presenting an uncontrolled hypertension, a pheochromocytoma, a carcinoid syndrome, a hyperthyroidism, a bipolar depression, a dysthymic schizophrenia, an acute confusional state, pophyria or a history of retrobulbar optic neuritis.
20. Patient who is participating or has participated in a clinical trial in the month prior to the study screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | 12 months after the end of treatment
  Clinical cure rate in the modified intent-to-treat (mITT)population during the hospital visit. Patients will be declared cured if clinical signs of infection are normalized.

SECONDARY OUTCOMES:
Cure rate | 12 months after the end of treatment
  Cure rate ine the modified intent-to-treat population during the hospital visit. Patients will be cdeclared cured if radiological and laboratory signs of infection are normalized.
Cure rate | 6 and 24 months after the end of treatment for the modified intent-to-treat population and at 12 months for the per protocol population.
  Patients will be declared cured if clinical, radiological, and laboratory signs of infection normalized.

CONTACTS AND LOCATIONS:
Overall Officials: Louis BERNARD, Principal Investigator — CHRU de Tours FRANCE; David BOUTOILLE, Principal Investigator — CHU de Nantes FRANCE; Gwenael LE MOAL, Principal Investigator — CHU de Poitiers FRANCE; Matteo BASSETTI, Principal Investigator — Azienda Opedaliera Universitaria San Maria della Misericordia ITALY; Silvano ESPOSITO, Principal Investigator — Facolta di Medicina e Chirugia ITALY; Jeannot GAUDIAS, Principal Investigator — Centre de Chirurgie Orthopédique et de la Main FRANCE; Alex SORIANO, Principal Investigator — Hospital Clinic of Barcelona SPAIN; Bartolome LLADO FERRER, Principal Investigator — Hospital Son Llatzer Palma Balears SPAIN; Mar SANCHEZ SOMOLINOS, Principal Investigator — HGU Gregorio Maranon Madrid SPAIN; Eric SENNEVILLE, Principal Investigator — CH de Tourcoing FRANCE
Locations (9):
- France (5):
  - CHRU de Tours, Tours, Indre et Loire
  - CHU de Nantes, Nantes
  - CHU de Poitiers, Poitiers
  - Centre de Chirurgie Orthopédique et de la Main, Strasbourg
  - CH de Tourcoing, Tourcoing
- Azienda Opedaliera Universitaria San Maria della Misericordia, Udine, Italy
- Spain (3):
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Son Llatzer, Palma de Mallorca